CLINICAL TRIAL: NCT02318056
Title: The Burn Glove Trial-A Randomized Controlled Trial of Dressings for Partial Thickness Hand Burns
Brief Title: The Burn Glove Trial - Hand Burn Dressing Pilot
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to reorganization.
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ABR-SIUSOM-14-002
Record Dates: First submitted 2014-07-23; First posted 2014-12-17 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Burns
Keywords: hand; burns; thermal; dressing; Aquacel®; Mepilex® Transfer Ag; Xeroform®; Bacitracin®; partial thickness; epithelialization; wound healing; scar; scarring
MeSH Terms: conditions — Burns; Cicatrix | interventions — Anti-Bacterial Agents; Bacitracin; 2,4,6-tribromophenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aquacel® Ag Burn Glove (Experimental): Application of Aquacel® Ag Burn Glove burn dressing
  Interventions: Other: Aquacel® Ag Burn Glove
- Mepilex® Transfer Ag (Active Comparator): Application of Mepilex® Transfer Ag burn dressing
  Interventions: Other: Mepilex® Transfer Ag
- Xeroform®/Bacitracin® (Active Comparator): Application of Xeroform® burn dressing and Bacitracin® topical antibiotic
  Interventions: Drug: antibiotic

INTERVENTIONS:
Other: Aquacel® Ag Burn Glove — burn dressing
  Other Names: ConvaTec
  Arms: Aquacel® Ag Burn Glove
Other: Mepilex® Transfer Ag — burn dressing
  Other Names: Safetac®; Molnlycke® Health Care
  Arms: Mepilex® Transfer Ag
Drug: antibiotic — antibiotic burn dressing
  Other Names: Bacitracin®; Xeroform®
  Arms: Xeroform®/Bacitracin®

SUMMARY:
Specific Aim 1: To determine if one of three burn dressings provides a less painful healing experience for partial thickness hand.

Specific Aim 2: To evaluate if one of three dressings provides greater functionality during and after healing of partial thickness hand burns.

Specific Aim 3: To determine if one of three burn dressings promotes aesthetically superior healing results for partial thickness hand burns.

DETAILED DESCRIPTION:
Various products are on the market and available for use on partial thickness burns to the hand/s. Our current institutional standard of care is to use Xeroform Gauze (Coviden, Mansfield, MA) and Bacitracin Ointment (Fougera, Melville, NY) to promote a moist antibacterial healing environment with the ability to monitor the healing progress daily. However, silver (AG) based dressings that employ nanocrystalline technology with hydrofiber (Aquacel AG burn; ConvaTec, Princeton, NJ) or soft silicone foam (Mepilex AG ; Molnlycke Health Care, Dunstable, United Kingdom) have been well accepted as alternative dressing solutions. These dressings have longer interval times between changes, leading to a reported increase in patient comfort, diminished skin shearing/stripping, and rapid re-epithelialization.

Given the anatomic intricacies, partial thickness burns to the hand present a challenge in dressing selection. Recently, ConvaTec unveiled the Aquacel AG Burn Glove for use on partial thickness hand burns. In line with this idea, our institution has now begun to fashion a novel burn glove out of Mepilex Transfer AG with good success. To date there are no known studies that compare Xeroform/Bacitracin, Aquacel AG burn glove or Mepilex Transfer AG dressing. The goal of this study is to compare these three burn dressings used to treat partial-thickness hand burns and their impact on pain, function, and aesthetic outcomes. We will also explore psychosocial issues related to hand burn dressing changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting at Memorial Medical or Southern Illinois University (SIU) Health Care
* Patients with partial-thickness burn injuries to the dorsum and/or palm of the hand/s that exceeds ½% total body surface area (TBSA) for at least one hand.
* < 10% TBSA 2nd and 3rd degree burn injuries
* Initial clinical presentation < 5 days post burn injury

Exclusion Criteria:

* < ½ % TBSA involving the hand
* > 10%TBSA burn injuries
* > 60 years of age
* < 8 years of age
* Patients (or parents of minors) without cognitive capacity to comprehend informed consent
* Presentation > 5 days post-burn injury event
* Pregnant women
* Full thickness/3rd degree burns to the dorsal and/or palmer hand/s
* Exposed vital structures (tendons, nerves, bone, vessels)
* Uncontrolled Type II Diabetes
* Type I Diabetes
* History of Chronic Obstructive Pulmonary Disease
* Have a known allergy to silver products
* Signs of infection on initial clinical presentation (presence of purulent drainage, significant cellulitis, and/or fever)
* Smoke/inhalation injuries requiring ventilation
* Critically ill patients requiring intensive care

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
pain | baseline to 6 months post-burn injury
  pain as measured by the Patient and Provider Scar Assessment Scale

SECONDARY OUTCOMES:
pain | baseline to 6 months post-burn injury
  pain as measured by the Michigan Hand Outcomes Questionnaire (MHQ)
pain | baseline to 6 months post-burn injury
  pain as measured by the Disabilities of the Arm, Shoulder and Hand Scale, Quick (QuickDASH)
functionality | baseline to 6 months post-burn injury
  functionality as measured by the Michigan Hand Outcomes Questionnaire (MHQ)
functionality | baseline to 6 months post-burn injury
  functionality as measured by the Disabilities of the Arm, Shoulder and Hand Scale, Quick (QuickDASH)
aesthetic appearance | baseline to 6 months post-burn injury
  scar formation and aesthetic appearance measured using the Vancouver Scar Scale
aesthetic appearance | baseline to 6 months post-burn injury
  scar formation and aesthetic appearance measured using the the Patient and Provider Scar Assessment Scale

OTHER OUTCOMES:
quality of life | baseline to 6 months post-burn injury
  quality of life measured by the psychosocial scales: Burn Specific Health Scale (BSHS)
resilience | baseline to 6 months post-burn injury
  resilience measured by the Connor-Davidson Resilience Scale (CD-RISC)

CONTACTS AND LOCATIONS:
Overall Officials: Nada N Berry, MD, Principal Investigator — Southern Illinois University
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wasiak J, Cleland H, Campbell F. Dressings for superficial and partial thickness burns. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD002106. doi: 10.1002/14651858.CD002106.pub3. PMID 18843629
- [Background] Robson MC, Smith DJ Jr, VanderZee AJ, Roberts L. Making the burned hand functional. Clin Plast Surg. 1992 Jul;19(3):663-71. PMID 1633673
- [Background] Kamolz LP, Kitzinger HB, Karle B, Frey M. The treatment of hand burns. Burns. 2009 May;35(3):327-37. doi: 10.1016/j.burns.2008.08.004. Epub 2008 Oct 25. PMID 18952379
- [Background] Walburn J, Vedhara K, Hankins M, Rixon L, Weinman J. Psychological stress and wound healing in humans: a systematic review and meta-analysis. J Psychosom Res. 2009 Sep;67(3):253-71. doi: 10.1016/j.jpsychores.2009.04.002. Epub 2009 Jul 2. PMID 19686881
- [Background] Atiyeh BS, Costagliola M, Hayek SN, Dibo SA. Effect of silver on burn wound infection control and healing: review of the literature. Burns. 2007 Mar;33(2):139-48. doi: 10.1016/j.burns.2006.06.010. Epub 2006 Nov 29. PMID 17137719
- [Background] Hollinger MA. Toxicological aspects of topical silver pharmaceuticals. Crit Rev Toxicol. 1996 May;26(3):255-60. doi: 10.3109/10408449609012524. PMID 8726163
- [Background] Bowler PG, Jones SA, Walker M, Parsons D. Microbicidal properties of a silver-containing hydrofiber dressing against a variety of burn wound pathogens. J Burn Care Rehabil. 2004 Mar-Apr;25(2):192-6. doi: 10.1097/01.bcr.0000112331.72232.1b. PMID 15091147
- See also: Institute for Plastic Surgery, Office for Clinical Research — http://www.siumed.edu/surgery/plastics/clinical-research.html